CLINICAL TRIAL: NCT04257864
Title: Impact of Bevacizumab Versus Docetaxel/Erlotinib on Tumor Metrics in Patients With Previously Untreated Advanced Non Small Cell Lung Cancer: A Study by the Hellenic Co-operative Oncology Group
Brief Title: Bevacizumab Versus Docetaxel/Erlotinib on Tumor Metrics in Patients With Previously Untreated Advanced Non Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: Neo-Doperlo
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Erlotinib followed by docetaxel: Erlotinib given for twelve consecutive days before docetaxel
- Docetaxel followed by erlotinib: Erlotinib given for twelve consecutive days after docetaxel
- Bevacizumab treated: Bevacizumab treated patients

SUMMARY:
To determine the more effective dosing sequence of intermittent erlotinib and docetaxel for treating patients with the diagnosis of advanced Non-Small-Lung-Cancer.

DETAILED DESCRIPTION:
In 2008, the Hellenic Co-operative Oncology group (HeCOG) initiated a randomized phase II study to determine the comparative efficacy of intermittent docetaxel/erlotinib chemotherapy, with erlotinib given for twelve consecutive days either before (group A) or after (group B) docetaxel, in chemotherapy-naive patients with advanced non small cell lung cancer. Docetaxel chemotherapy was considered one of the valid non-platinum containing therapeutic options at that time and today represents one of the approved second-line treatment options after failure of first-line platinum based chemotherapy. The trial was terminated early due to slow accrual after enrollment of 51 patients and was published in 2014, showing no clinically meaningful difference between the two treatment arms.

Based on the aforementioned trial population,a parallel radiological study was conducted, evaluating sequential tumor metrics on computed tomography performed at baseline and after each cycle of treatment in patients receiving either bevacizumab or docetaxel/erlotinib. Given the differential mechanism of action of these agents, it was hypothesized that the different parameters of radiological tumor response evaluation, namely the maximum diameter, tumor volume and tumor density, would respond differently for each therapeutic category (a chemotherapeutic agent, a molecular agent and and an anti-angiogenic agent). For bevacizumab, in particular, it was hypothesized that its unique mechanism of action, inducing central tumor necrosis and subsequent shrinkage, would lead to completely different tumor metrics as compared to the other two agents. Herein the final results of this analysis are presented, showing the comparison of the three agents in terms of tumor response metrics, as evaluated in CT scans performed at baseline and after each cycle of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 75 years inclusive, with histologically confirmed metastatic non small cell lung cancer will be enrolled.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
3. Presence of measurable or evaluable disease (lesions that are present but do not fulfil the criteria for measurable disease).

Exclusion Criteria:

1. Patients who have undergone complete tumor resection after responding to platinum based chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non small cell lung cancer evaluated with Computed Scan or Magnetic Resonance Imaging.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Tumor response | Every 12 -16 weeks
  Evaluation of response using RECIST 1.1 criteria (REF) was based on the measurement of a total of 5 measurable lesions.